CLINICAL TRIAL: NCT06694376
Title: Understanding and Expanding the Reach of Home Visiting (HV-REACH) Project
Acronym: HV-REACH
Status: Not yet recruiting | Type: Observational
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Brazelton Touchpoints Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: MPR51320; 47QRAA18D00BQ/75ACF121F80023 (Other Grant/Funding Number: U.S. DHHS, ACF, OPRE)
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Home Visiting; Centralized Intake Systems
Keywords: Home visiting; MIECHV; Early care and education; Centralized intake systems

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single-group study: The study has one group/cohort, which will include up to 154 people. The study team will conduct one round of semi-structured interviews with up to 42 administrators or other staff at the centralized intake system organization(s), 28 home visiting program directors and other staff responsible for overseeing outreach and enrollment, 42 home visitors and other staff responsible for conducting outreach and enrollment, and 42 families who were referred to home visiting through the selected centralized intake systems. All respondents will also complete a form to provide information about their demographic characteristics.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention.

SUMMARY:
Mathematica, funded by the Administration for Children and Families (ACF) Office of Planning, Research, and Evaluation (OPRE) in the U.S. Department of Health and Human Services (HHS) will collect descriptive information for the Understanding and Expanding the Reach of Home Visiting (HV-REACH) project. The study team will conduct qualitative case studies in up to seven purposively selected centralized intake systems that refer families to Early Childhood Home Visiting programs. Centralized intake systems are a single entry point that use outreach and screening to identify families with needs and provide referrals to the home visiting program that best fits those needs. Existing centralized intake systems use a range of methods, and their definitions and applications can vary widely.

The goal of the case studies is to provide an in-depth understanding of the features of centralized intake systems, how they reach potentially eligible families, and how they support and expand the enrollment of families in early childhood home visiting (ECHV) programs. Understanding and explaining how staff think different features of these systems influence family and staff experiences of outreach, screening, referral, and enrollment processes can potentially lead to opportunities for program improvement efforts, technical assistance, or changes to centralized intake system processes. For instance, ACF and their partner, the Health Resources and Services Administration (HRSA), can use information about different centralized intake systems to develop policy and program guidance. In addition, the public-including current centralized intake systems, staff from localities considering implementing them, and technical assistance providers who work with centralized intake systems-can use information from the case studies about (1) successfully implementing or enhancing existing centralized intake systems, or (2) utilizing new outreach or referral pathways to expand enrollment to families not consistently reached. For example, staff from localities considering implementing centralized intake systems can understand different staffing and governance structures that might work in their contexts. Researchers can also use the information to plan future studies of centralized intake systems that examine the outcomes of these systems.

Data collection will begin in fall 2024. The study team will conduct virtual or in-person site visits, with semi-structured interviews and document collection, to understand different features of these systems and family and staff experiences with outreach, screening, referrals, and enrollment processes.

DETAILED DESCRIPTION:
The Maternal, Infant, and Early Childhood Home Visiting (MIECHV) Program, an evidence-based service delivery model, can support child and maternal health, child development and school readiness, and family economic self-sufficiency, and help reduce child abuse and neglect. Early childhood home visiting (ECHV) programs collectively reached about 278,000 families in the United States in 2021, while MIECHV-funded programs reached about 71,000 families (Health Resources and Services Administration [HRSA], 2022; National Home Visiting Resource Center [NHVRC], 2022). However, many more families are eligible for and could benefit from these programs. In conducting the Understanding and Expanding the Reach of Home Visiting (HV-REACH) project, the Administration for Children and Families (ACF) aims to deepen understanding of how home visiting can better reach families, including: (1) families who are not recruited in the first place; (2) families who are recruited for home visiting but do not enroll; (3) families who enroll, but never engage to receive services; and (4) families who are recruited and engage initially, but end their participation early.

By streamlining screening and referral processes, centralized intake systems may help improve enrollment of families across different referral pathways. These types of systems have been in existence for decades and have become increasingly widespread in recent years (National Evidence-Based Home Visiting Model Alliance [NHVMA], 2018; Roberts et al., 1996). However, no studies have systemically documented the various types of systems. In addition, the ways in which home visiting programs interact with the systems and the influence these systems have on family experiences around outreach, screening, referrals, and enrollment-particularly for those that are underserved or may be missed by a system's referral pathways-is largely unknown.

The HV-REACH project will conduct qualitative case studies to provide an in-depth understanding of the features of centralized intake systems, how they reach potentially eligible families, and how they support and expand the enrollment of families in ECHV programs. To carry out the case studies, the HV-REACH study team will conduct virtual or in-person site visits in up to seven sites. A site includes an organization or organizations that run a selected centralized intake system and one or two associated home visiting programs that receive referrals from the selected centralized intake system. The study team defines a home visiting program as an organization that delivers ECHV services. The study team will purposively select up to seven sites that fall into different models of identified centralized intake systems-for example, triage model, shared decision-making, and market (NHVMA, 2018). Recruitment will cease after seven sites agree to participate.

Each site visit will include one round of semi-structured interviews with administrators or other staff at the centralized intake system organization(s) (up to 6 respondents per site), home visiting program directors and other staff responsible for overseeing outreach and enrollment (up to 4 respondents per site from up to two different home visiting programs), home visitors and other staff responsible for conducting outreach and enrollment (up to 6 respondents in up to 4 interviews per site), and families who were referred to home visiting through the selected centralized intake systems (up to 6 respondents per site). The study team will purposively select respondents to provide a range of perspectives on the study's research questions.

The results are not intended to promote statistical generalization to different sites or service populations beyond the sample. The research team does not intend for this information to be used as the principal basis for public policy decisions.

ELIGIBILITY:
Inclusion Criteria:

* Centralized intake administrator or other staff at selected centralized intake system organization
* Program director at home visiting program or other staff responsible for overseeing outreach and enrollment at home visiting program associated with selected centralized intake system
* Home visitor at home visiting program or other staff responsible for conducting outreach and enrollment at home visiting program associated with selected centralized intake system
* Families referred to home visiting through selected centralized intake system at home visiting program associated with selected centralized intake system

Exclusion Criteria:

* Does not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample. From the seven selected sites: centralized intake administrators and other staff at centralized intake system organization, home visiting program directors or other staff responsible for overseeing outreach and enrollment, home visitor at home visiting program or other staff responsible for conducting outreach and enrollment, and families who are referred to home visiting through the centralized intake system.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-08-29 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Centralized Intake Administrator Screening Talking Points or Screening Email with Questions | 2 months
  Study-developed email outreach will gather information about whether a nominated centralized intake system organization is eligible to participate in the study.
Centralized Intake Administrator and Other Staff Interview Protocol | 5 months
  Study-developed interview protocol will learn from centralized intake administrators and other staff about how centralized intake systems operate; how they coordinate with home visiting programs to screen, refer, and enroll families for home visiting programs; and about opportunities to improve staff or family experience with centralized intake systems.
Document Review Request | 5 months
  Study-developed document review request will be used to gather documents through which we will learn about types of materials and documentation that centralized intake systems use related to outreach, screening, referrals, and enrollment processes and pathways.
Home Visiting Program Director and Other Staff Interview Protocol | 5 months
  Study-developed interview protocol will learn from home visiting program directors and other staff about how centralized intake systems operate; how they coordinate with centralized intake systems to screen, refer, and enroll families for home visiting programs; and about opportunities to improve staff or family experience with centralized intake systems.
Home Visitor and Other Staff Interview Protocol | 5 months
  Study-developed interview protocol will learn about how home visitors contribute to and support family referral and enrollment processes, and about opportunities to improve the home visitor or family experience with centralized intake systems.
Family Interview Protocol | 5 months
  Study-developed interview protocol will learn about experiences of parents or caregivers, and perceptions of centralized intake systems in terms of eligibility, wait times, referrals, communication, and relationships with centralized intake or home visiting program staff.
Participant Characteristics Form | 5 months
  Study-developed survey instrument will collect information about centralized intake administrators', home visiting program directors', home visitors', and parent/caregivers' race and/or ethnicity, age, and gender identity. We will also ask parent/caregivers to provide information to provide information about number of children, child ages, and primary language. Responses will be anonymous.

CONTACTS AND LOCATIONS:
Locations (1):
- Mathematica, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Information about respondents will be kept private to the extent permitted by law. Any data shared for the project will be shared in summary form. Data that are collected will be destroyed when the study concludes.

REFERENCES:
- [Background] Roberts, R. N., Akers, A. L., & Behl, D. D. (1996). Family-level service coordination within home visiting programs." Topics in Early Childhood Special Education, 16(3), 279-301. https://doi.org/10.1177/027112149601600303.
- See also: Provides information cited in Detailed Description section — https://mchb.hrsa.gov/sites/default/files/mchb/about-us/program-brief.pdf
- See also: Provides information cited in Detailed Description section — https://www.nationalalliancehvmodels.org/_files/ugd/bc26e2_389831a76eaa41eaba7bb2b376a47816.pdf
- See also: Provides information cited in Detailed Description section — https://nhvrc.org/yearbook/2022-yearbook/